CLINICAL TRIAL: NCT00221325
Title: Phase I Study of Intraventricular Administration of Rituximab in Combination With Methotrexate in the Treatment of Recurrent CNS and Intraocular Lymphoma
Brief Title: A Safety Study of Rituximab Plus MTX Injected Into the Cerebrospinal Fluid in the Treatment of Brain Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC05254; H9414-29670
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Central Nervous System Lymphoma; Intraocular Lymphoma
Keywords: Phase I Clinical Trial; Pharmacokinetics; Pharmacodynamics; CNS Lymphoma; Ocular Lymphoma
MeSH Terms: conditions — Intraocular Lymphoma | interventions — Methotrexate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab Plus MTX (Experimental)
  Interventions: Drug: Intraventricular Rituximab Plus MTX

INTERVENTIONS:
Drug: Intraventricular Rituximab Plus MTX — Intraventricular injection of rituximab into an Ommaya reservoir on day 1 of each week. Intraventricular rituximab plus methotrexate (MTX) on day 4 of each week.
  First three patients at dose A : 25 mg rituximab on day 1, and MTX (12 mg) plus rituximab (10 mg) on day 4 each week.
  If there are no dose limiting toxicities at Dose A in all of the first 3 patients or in 5 of the first 6 patients, the next 3 patients will receive dose level B: 25 mg rituximab on day 1, and combination MTX (12 mg) plus rituximab (25 mg) on day 4 of each week.
  Oral leucovorin rescue 24 hours after each MTX administration. Maximum injections will be 16 over 9-weeks. Subjects who experience a partial response at week 10 will be given the option for extended dosing.
  Other Names: MTX; amethopterin; Rituxan; MabThera

SUMMARY:
Rituximab is the first monoclonal antibody to receive approval in the treatment of cancer and has been proven to lead to extended survival when administered intravenously in the treatment of patients with systemic non-Hodgkin's lymphoma. We have previously demonstrated that a small fraction of Rituximab administered intravenously is able to cross the blood-brain-barrier into the brain.

We will test the idea that the direct injection into the cerebrospinal fluid of Rituximab, a monoclonal antibody which attacks and kills lymphoma cells, is safe and when used in combination with methotrexate in patients with recurrent brain and intraocular lymphoma.

We will also test the idea that the combination of rituximab plus methotrexate has activity and is effective in the treatment of recurrent brain and intraocular lymphoma.

DETAILED DESCRIPTION:
Rituximab is the first monoclonal antibody to receive FDA approval in the treatment of cancer. Intravenous administration of rituximab has been demonstrated to lead to prolongation of survival when used in combination with chemotherapy in the treatment of patients with systemic non-Hodgkin's lymphoma. We have previously demonstrated that a small fraction of Rituximab administered intravenously is able to cross the blood-brain-barrier into the brain and we have also previously demonstrated that direct intraventricular administration of Rituximab is able to achieve high concentrations within the cerebrospinal fluid ventricles and lumbar sac.

We will test the hypothesis that the direct intraventricular injection of Rituximab in combination with Methotrexate is safe and when used in combination in patients with recurrent brain and intraocular lymphoma. We will evaluate the safety of this combination by testing different dose levels of Rituximab. We will also measure the concentration of Rituximab in the intraocular compartments and cerebrospinal fluid at different time points after intraventricular administration to determine the pharmacokinetics of intrathecal Rituximab as well as the potential impact of Methotrexate on Rituximab distribution.

We will also test the hypothesis that the intraventricular administration of the combination of rituximab plus methotrexate has activity and is effective in the treatment of recurrent brain and intraocular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed, refractory CNS lymphoma, ocular lymphoma, lymphomatous meningitis
2. Tumors must be CD20 + on pathologic analysis.
3. Patients must have an Ommaya reservoir (ventricular access device.
4. Patients may have had prior intrathecal methotrexate, ara-C or thiotepa but must have recovered from any reversible toxicity caused by prior treatment.
5. Concurrent systemic chemotherapy is allowed for treatment of disease outside the meninges with the exception of high-dose methotrexate (>500 mg/m2/d, high-dose ara-C (> 2 gm/m2/d), high-dose thiotepa (>300 mg/m2/d) or investigational agents.
6. Patients must have sufficient baseline hematologic function: >1,500 granulocytes and >50,000 platelets/ul.
7. Patients must have had a nuclear medicine CSF flow study performed within 30 days of treatment which shows no significant obstruction within the ventricles.

Exclusion Criteria:

1. History of whole brain or craniospinal irradiation or intrathecal chemotherapy < 4 days before initiation of intra-CSF administration of rituximab.
2. Anticipated survival of less than one month.
3. HIV infection. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-04; Primary Completion 2012-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
whether intra-CSF administration of rituximab in combination with MTX in patients with recurrent CNS and intraocular lymphoma is associated with neurotoxicity | 4 weeks

SECONDARY OUTCOMES:
To define the rate of tumor response (CR plus PR) in the brain, spine, eye, or CSF. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James L. Rubenstein, MD PhD, Study Chair — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Rubenstein JL, Li J, Chen L, Advani R, Drappatz J, Gerstner E, Batchelor T, Krouwer H, Hwang J, Auerback G, Kadoch C, Lowell C, Munster P, Cha S, Shuman MA, Damon LE. Multicenter phase 1 trial of intraventricular immunochemotherapy in recurrent CNS lymphoma. Blood. 2013 Jan 31;121(5):745-51. doi: 10.1182/blood-2012-07-440974. Epub 2012 Nov 29. PMID 23197589